CLINICAL TRIAL: NCT03226457
Title: Renal and Cardiovascular Effect of Sodium-Glucose Co-Transporter 2 (SGLT2) Inhibition in Combination With Loop Diuretics in Diabetic Patients With Chronic Heart Failure
Brief Title: SGLT2 Inhibition in Combination With Diuretics in Heart Failure
Acronym: RECEDE-CHF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Dundee (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Principal Investigator, Natalie Mordi, British Heart Foundation Clinical Research Fellow, University of Dundee
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BHF:807998
Record Dates: First submitted 2017-07-17; First posted 2017-07-21 (Actual); Results first posted 2021-06-30 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Heart Failure; Type 2 Diabetes Mellitus
Keywords: Heart Failure; Type 2 Diabetes Mellitus; Sodium-Glucose co-Transporter 2 (SGLT2) inhibitors; Natriuresis; Diuresis
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus, Type 2 | interventions — empagliflozin; Furosemide

STUDY DESIGN:
Intervention Model Description: 6 week period of Investigational Medicinal Product (Empagliflozin 25 mg od) or placebo. A 2 week washout period will then be observed, followed by the second arm with a further 6 week period of placebo or IMP. At week 1 and week 6 of each arm, detailed Renal Physiology Test days will be performed.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Empagliflozin/Placebo (Active Comparator): Empagliflozin (SGLT2 inhibitor) 25mg capsules once daily for 6 weeks, minimum of a 2 week washout period, then 6 weeks placebo
  Interventions: Drug: Empagliflozin 25mg; Drug: Placebo oral capsule; Drug: Frusemide
- Placebo/Empagliflozin (Active Comparator): Placebo for 6 weeks, minimum of a 2 week washout period, followed by Empagliflozin (SGLT2 inhibitor) 25mg capsules once daily for 6 weeks
  Interventions: Drug: Empagliflozin 25mg; Drug: Placebo oral capsule; Drug: Frusemide

INTERVENTIONS:
Drug: Empagliflozin 25mg — Empagliflozin (SGLT2 inhibitor) 25 mg once daily for 6 weeks
  Other Names: Jardiance
Drug: Placebo oral capsule — Capsules containing microcrystalline cellulose Ph Eur over encapsulated in a hard gelatine capsule shell to match the active comparator once daily for 6 weeks
  Other Names: Placebo
Drug: Frusemide — Renal Physiology Test (RPT) days will be performed at week 1 and week 6 on each arm of this crossover trial. On these RPT days participants will undergo oral water loading (15mls/kg) and frequent urination at 30 minute intervals to gain a steady state diuresis. At a set time point, an intravenous bolus of furosemide at a dose of half the participant's usual loop diuretic dose will be administered.

SUMMARY:
The RECEDE-CHF trial is a single centre phase IV, randomised, double-blind, placebo-controlled, crossover trial conducted in NHS Tayside, Scotland comparing empagliflozin 25mg, to placebo in patients with Type 2 Diabetes and mild Chronic Heart Failure with left ventricular systolic dysfunction who are already on a loop diuretic. Renal physiological testing will be performed at two points on each arm to assess the effect of empagliflozin, on urinary volume, compared to placebo. The secondary outcomes are to assess the effect of empagliflozin in addition to loop diuretics on natriuresis, to assess the safety of add-on SGLT2 inhibitor therapy as measured by changes to serum creatinine and eGFR, to assess effects of empagliflozin on urinary protein/creatinine ratio, albumin/creatinine ratio and cystatin C when compared to placebo.

DETAILED DESCRIPTION:
Type 2 Diabetes (T2D) and Heart Failure (HF) are a frequent combination, where treatment options remain limited. There has been increasing interest around the sodium-glucose co-transporter 2 (SGLT2) inhibitors and their use in patients with HF. This is following publication of EMPA-REG OUTCOME trial that reported a 14% reduction in the primary composite outcome of cardiovascular death, non-fatal myocardial infarction, non-fatal stroke and >30% reductions in cardiovascular mortality, overall mortality and HF hospitalisations in patients randomised to the SGLT2 inhibitor, empagliflozin, when compared to placebo. Data on the effect of SGLT2 inhibitor use with diuretics is limited. We hypothesize that, in the diabetic CHF population, SGLT2 inhibition may augment the effects of loop diuretics.

Renal Physiology Test (RPT) days will be performed at week 1 and week 6 on each arm of this crossover trial. On these RPT days participants will undergo oral water loading (15mls/kg) and frequent urination at 30 minute intervals to gain a steady state diuresis. The investigational medicinal product will be administered, followed by an intravenous bolus of furosemide at a dose of half the participant's usual loop diuretic dose.

This proof of concept trial will aim to shed light on the mechanism of the cardiovascular and renal outcomes demonstrated in the recent EMPA-REG study by documenting the influence of the SGLT2 inhibitors when used in combination with a loop diuretic on diuresis and natriuresis when compared to placebo.

The RECEDE-CHF trial is funded by the British Heart Foundation (BHF grant number: 807998). NAM is a BHF funded clinical research fellow.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of NYHA Functional class II-III HF with prior echocardiographic evidence of LVSD.
* On stable doses of furosemide, or alternative loop diuretic for at least one month.
* Stable Type 2 Diabetes (HbA1c, in the last 3 months, of 6.5% ≤ and ≤10.0%)
* eGFR ≥ 45 ml/min.
* Have stable HF symptoms for at least three months prior to consent
* On stable HF therapy for at least three months prior to consent
* Have not been hospitalised for HF for at least three months prior to consent.
* Women of childbearing potential must agree to take precautions to avoid pregnancy throughout the trial and for 4 weeks after intake of the last dose.

Exclusion Criteria:

* A diagnosis of chronic liver disease and/or liver enzymes that are twice the upper limit of normal
* Systolic BP of <95mmHg at screening visit.
* Participants on thiazide diuretics.
* Participants receiving renal dialysis
* Participants who have previously had an episode of diabetic ketoacidosis.
* Participants with type 1 diabetes mellitus
* Malignancy (receiving active treatment) or other life threatening disease.
* Pregnant or lactating women
* Participants with difficulty in micturition e.g. severe prostate enlargement
* Allergy to any SGLT2 inhibitor or lactose or galactose intolerance
* Past or current treatment with any SGLT2 inhibitor
* Participants who have participated in any other clinical interventional trial of an investigational medicinal product within 30 days.
* Participants who are unable to give informed consent
* Any other reason considered by the physician to be inappropriate for inclusion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2018-12-11 (Actual); Study Completion 2019-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natalie A Mordi, MBChB MRCP, Principal Investigator — University of Dundee
Locations (1):
- University of Dundee, Ninewells Hospital and Medical School, Dundee, Angus, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mordi NA, Mordi IR, Singh JS, McCrimmon RJ, Struthers AD, Lang CC. Renal and Cardiovascular Effects of SGLT2 Inhibition in Combination With Loop Diuretics in Patients With Type 2 Diabetes and Chronic Heart Failure: The RECEDE-CHF Trial. Circulation. 2020 Nov 3;142(18):1713-1724. doi: 10.1161/CIRCULATIONAHA.120.048739. Epub 2020 Aug 29. PMID 32865004
- [Derived] Mordi NA, Mordi IR, Singh JS, Baig F, Choy AM, McCrimmon RJ, Struthers AD, Lang CC. Renal and Cardiovascular Effects of sodium-glucose cotransporter 2 (SGLT2) inhibition in combination with loop Diuretics in diabetic patients with Chronic Heart Failure (RECEDE-CHF): protocol for a randomised controlled double-blind cross-over trial. BMJ Open. 2017 Oct 16;7(10):e018097. doi: 10.1136/bmjopen-2017-018097. PMID 29042392

RESULTS

PARTICIPANT FLOW:
Groups:
- Empagliflozin/Placebo: Treatment Sequence:
  Empagliflozin (SGLT2 inhibitor) 25mg capsules once daily for 6 weeks
  Empagliflozin 25mg: Empagliflozin (SGLT2 inhibitor) 25 mg once daily for 6 weeks
  Frusemide: Renal Physiology Test (RPT) days will be performed at week 1 and week 6 on each arm of this crossover trial. On these RPT days participants will undergo oral water loading (15mls/kg) and frequent urination at 30 minute intervals to gain a steady state diuresis. At a set time point, an intravenous bolus of furosemide at a dose of half the participant's usual loop diuretic dose will be administered.
  Minimum of a 2 week washout period.
  6 weeks of placebo
- Placebo/Empagliflozin: Treatment Sequence:
  Capsules containing microcrystalline cellulose Ph Eur over encapsulated in a hard gelatine capsule shell to match the active comparator
  Placebo oral capsule: Capsules containing microcrystalline cellulose Ph Eur over encapsulated in a hard gelatine capsule shell to match the active comparator once daily for 6 weeks
  Frusemide: Renal Physiology Test (RPT) days will be performed at week 1 and week 6 on each arm of this crossover trial. On these RPT days participants will undergo oral water loading (15mls/kg) and frequent urination at 30 minute intervals to gain a steady state diuresis. At a set time point, an intravenous bolus of furosemide at a dose of half the participant's usual loop diuretic dose will be administered.
  Minimum of 2 week washout period
  6 weeks of Empagliflozin 25mg: Empagliflozin (SGLT2 inhibitor) 25 mg once daily
Period: Treatment 1: 6 Weeks
Arm/Group | Empagliflozin/Placebo | Placebo/Empagliflozin
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0
Period: Washout Period: Minimum 2 Weeks
Arm/Group | Empagliflozin/Placebo | Placebo/Empagliflozin
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0
Period: Treatment 2: 6 Weeks
Arm/Group | Empagliflozin/Placebo | Placebo/Empagliflozin
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Baseline Characteristics: N = 23, Crossover study design. Baseline characteristics
Arm/Group | Baseline Characteristics
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.8 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 23

OUTCOME MEASURES:

1. Primary Outcome: The Effect of Empagliflozin Versus Placebo on the Change in Urine Output.
Description: Change from urinary volume from baseline (mls).
Time Frame: Change from baseline to 6 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: mL
Groups:
- Empagliflozin: Empagliflozin (SGLT2 inhibitor) 25mg capsules once daily for 6 weeks
  Empagliflozin 25mg: Empagliflozin (SGLT2 inhibitor) 25 mg once daily for 6 weeks
  Frusemide: Renal Physiology Test (RPT) days will be performed at week 1 and week 6 on each arm of this crossover trial. On these RPT days participants will undergo oral water loading (15mls/kg) and frequent urination at 30 minute intervals to gain a steady state diuresis. At a set time point, an intravenous bolus of furosemide at a dose of half the participant's usual loop diuretic dose will be administered.
- Placebo: Capsules containing microcrystalline cellulose Ph Eur over encapsulated in a hard gelatine capsule shell to match the active comparator
  Placebo oral capsule: Capsules containing microcrystalline cellulose Ph Eur over encapsulated in a hard gelatine capsule shell to match the active comparator once daily for 6 weeks
  Frusemide: Renal Physiology Test (RPT) days will be performed at week 1 and week 6 on each arm of this crossover trial. On these RPT days participants will undergo oral water loading (15mls/kg) and frequent urination at 30 minute intervals to gain a steady state diuresis. At a set time point, an intravenous bolus of furosemide at a dose of half the participant's usual loop diuretic dose will be administered.
Arm/Group | Empagliflozin | Placebo
Number analyzed (Participants) | 23 | 23
mL | 545 [136 to 954] | -113 [-345 to 119]
Statistical Analysis 1: Comparison: Empagliflozin vs Placebo; Details on the statistical analysis are published in the Circulation, DOI: 10.1161/CIRCULATIONAHA.120.048739 Analyses were performed on the primary and secondary measures comparing empagliflozin versus placebo and assessed by 2-way analysis of covariance correcting for treatment order, baseline value, and any percentage change in furosemide dose at the visit. Data for continuous outcome measures were assessed for normality before analysis; Test type: Other — Details of the power calculation are published in the Circulation, DOI: 10.1161/CIRCULATIONAHA.120.048739; p = 0.005, ANCOVA — (calculated)

2. Secondary Outcome: The Effect of Empagliflozin Versus Placebo on the Change in Urinary Sodium Excretion.
Description: The effect of empagliflozin versus placebo on the change in urinary sodium excretion: change in fractional urinary sodium excretion from baseline (%).
Time Frame: Change from baseline to 6 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of change in FENa
Arm/Group | Empagliflozin | Placebo
Number analyzed (Participants) | 23 | 23
percentage of change in FENa | 0.11 [-0.22 to 0.44] | -0.00 [-0.19 to 0.19]

3. Secondary Outcome: Number of Participants With a Change in CKD Category as Dictated by the Glomerular Filtration Rate
Description: The effect of empagliflozin versus placebo on the change in glomerular filtration rate: Change in estimated glomerular filtration rate from baseline (ml/min/1.73m2).
  Data was recorded as a persistent reduction in CKD category in the empagliflozin group versus placebo
Time Frame: From baseline to 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Empagliflozin | Placebo
Number analyzed (Participants) | 23 | 23
Participants | 6 | 5

4. Secondary Outcome: The Effect of Empagliflozin Versus Placebo on the Change in Serum Creatinine.
Description: Change in serum creatinine from baseline (mmol/L).
Time Frame: Change from baseline to 6 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Empagliflozin | Placebo
Number analyzed (Participants) | 23 | 23
mmol/L | -0.44 [-8.82 to 7.94] | -10.81 [-19.2 to -2.44]

5. Secondary Outcome: The Effect of Empagliflozin Versus Placebo on the Change to Urinary Protein/Creatinine Ratio.
Description: The effect of empagliflozin versus placebo on the change to urinary protein/creatinine ratio: Change in urinary protein/creatinine ratio from baseline (mg/mmol).
Time Frame: Change from baseline to 6 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/mmol
Arm/Group | Empagliflozin | Placebo
Number analyzed (Participants) | 12 | 11
mg/mmol | 2.26 [-1.75 to 6.28] | -3.05 [-7.05 to 0.97]

6. Secondary Outcome: The Effect of Empagliflozin Versus Placebo on the Change to Urinary Albumin/Creatinine Ratio.
Description: The effect of empagliflozin versus placebo on the change to urinary albumin/creatinine ratio: Change in urinary albumin/creatinine ratio from baseline (mg/mmol).
Time Frame: Change from baseline to 6 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/mmol
Arm/Group | Empagliflozin | Placebo
Number analyzed (Participants) | 23 | 23
mg/mmol | 1.18 [-0.69 to 3.05] | -1.1 [-2.98 to 0.77]

7. Secondary Outcome: The Effect of Empagliflozin Versus Placebo on the Change to the Renal Biomarker, Cystatin C.
Description: The effect of empagliflozin versus placebo on the change to the renal biomarker, cystatin C: Change in Cystatin C from baseline (ng/ml).
Time Frame: Change from baseline to 6 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: ng/ml
Arm/Group | Empagliflozin | Placebo
Number analyzed (Participants) | 23 | 23
ng/ml | 31.35 [-80.07 to 142.75] | 22.5 [-91.52 to 136.52]

ADVERSE EVENTS:
Time Frame: For the duration of the participants inclusion in the study to the point of completion e.g. 14 to 16 weeks in the trial, with a further review at 4 weeks following discontinuation of the investigational medicinal product e.g. 18 to 20 weeks in total.
Description: Because of the large volume of multicenter studies reporting on the safety and adverse events of SGLT2 inhibitors, for this trial the focus was on the effects on the coprescription with loop diuretic. Adverse event data were also collected.
  As a crossover study, the adverse event reporting is separated into the events that occurred on the specific intervention/treatment arms.
Arm/Group | Empagliflozin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 2/23 | 0/23
Other Adverse Events (participants affected / at risk) | 1/23 | 2/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Empagliflozin (N=23) | Placebo (N=23)
Hospitalization with heart failure following discontinuation of investigational medicinal product (Cardiac disorders) | 2 (2) | 0
Hypotension (Cardiac disorders) | 1 (1) | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Empagliflozin (N=23) | Placebo (N=23)
Gout (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) — Gout

LIMITATIONS AND CAVEATS:
Small, single-center crossover study. The dose investigated was 25mg empagliflozin, whereas in routine practice 10mg dose is most commonly used. We did not measure urine glucose in this study. Patients were only observed for 2 hours after administration of investigational medical. Any significant diuretic or natriuretic effect beyond this may have not been observed during this short time frame.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-01-22): https://cdn.clinicaltrials.gov/large-docs/57/NCT03226457/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-01): https://cdn.clinicaltrials.gov/large-docs/57/NCT03226457/SAP_001.pdf